CLINICAL TRIAL: NCT04790656
Title: Effects of Continuous Positive Airway Pressure (CPAP)and Physical Exercise on Cycle Ergometer in Myocardial Revascularization Post-surgical Patients
Brief Title: Interventional Effects on Myocardial Revascularization Post-surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00874 Arjumand Bano
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Myocardial Revascularization

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Therapy (Active Comparator): The control program will consist of progressive exercises according to each postoperative day. Two daily sessions with an average duration of 25 min will be performed. In addition to the physiotherapeutic program standardized by the hospital's team of physical therapists, the intervention group will perform physical exercise on a cycle ergometer with CPAP.
  Interventions: Other: Conventional Therapy
- Cycle ergometer combine with CPAP (Experimental): Physical exercise on a cycle ergometer combine with CPAP will be performed in a single daily session from the second to the fourth postoperative days
  Interventions: Other: Cycle ergometer combine with CPAP

INTERVENTIONS:
Other: Conventional Therapy — Subjects will randomly placed into intervention group and control group . In addition to the physiotherapeutic program standardized by the hospital's team of physical therapists, the intervention group will perform physical exercise on a cycle ergometer with CPAP.
  Arms: Conventional Therapy
Other: Cycle ergometer combine with CPAP — Physical exercise on a cycle ergometer combine with CPAP will be performed in a single daily session from the second to the fourth postoperative days . The maximum exercise time for postoperative day 2 will be 20 min, and 30 min for the third and fourth postoperative days.
  Arms: Cycle ergometer combine with CPAP

SUMMARY:
The aim is to evaluate the effectiveness of physical exercise on a cycle ergometer combine with CPAP in the postoperative period after myocardial revascularization

DETAILED DESCRIPTION:
Physical exercise on a cycle ergometer combine with CPAP as an adjunct to the rehabilitation of hospitalized subjects who will undergo myocardial revascularization will be safe, decrease the length of stay in the ICU, and help maintain functional capacity

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone myocardial revascularization surgery
* An ejection fraction of greater than40%
* Post operative mechanical ventilation for <12hours
* No definite diagnosis of chronic obstructive pulmonary disease and asthma

Exclusion Criteria:

* With complications in post operative period (e.g., Artial fibrillation, prolonged mechanical ventilation)
* Hemodynamically unstable patients
* Intolerance to CPAP(continuous positive airway)mask

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Modified Borg scale | 4th day
  The Modified Borg Dyspnoea Scale is most commonly used to assess symptoms of breathlessness. Despite being a subjective measure of exercise intensity, RPE scales provide valuable information when used correctly.
6 min walk distance | 4th day
  The six minute walking test (6MWT) was developed by the American Thoracic Society and it was officially introduced in 2002, coming along with a comprehensive guideline. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
1 min sit to stand test | 4th day
  Vaidya et al reported that 1-minute STS test is a simple and sensitive test and appears to be a practical, reliable, valid, and responsive alternative for measuring exercise capacity, particularly where space and time are limited
Digital Monovacumeter | 4th day
  The manovacuometer is a simple, quick and non-invasive test which measures the maximal respiratory pressures (MRS).Digital manovacuometer is a reliable and valid instrument for assessing maximum inspiratory pressure and maximum expiratory pressure in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- Rawalpindi institute of cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No